CLINICAL TRIAL: NCT00568607
Title: Phase II Study of a Combination Chemotherapy of DICE in the Patients With NK/T Cell Lymphoma
Brief Title: Study on the Combination Regimen of Dexamethasone Ifosfamide Cisplatin Etoposide in Patients With NK/T Cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Base for Drug Clinical Trials, Fudan University Cancer Hospital, Fudan University Cancer Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DICE-NK/T
Record Dates: First submitted 2007-12-05; First posted 2007-12-06 (Estimated); Last update posted 2010-09-08 (Estimated); Status verified 2010-09

CONDITIONS: Lymphoma
Keywords: NK/T cell lymphoma; Response Rate; TTP; OS; Toxicities
MeSH Terms: conditions — Lymphoma; Lymphoma, Extranodal NK-T-Cell | interventions — Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IFO, VP-16, DDP, DXM (Experimental)
  Interventions: Drug: IFO, VP-16, DDP, DXM

INTERVENTIONS:
Drug: IFO, VP-16, DDP, DXM — DXM 40 mg d1-4; IFO 1200mg/m2 d1-4; Mesna 400mg, tid, d1-4; VP-16 75 mg/m2 d1-4; DDP 20mg/m2 d1-4; q3w. Efficacy was evaluated every two cycles. If patients hadn't diseases progression, two more cycles and radiation would be administered.
  Other Names: DICE

SUMMARY:
The purpose of this study is to evaluate the efficacy and tolerability of the combination chemotherapy of DICE in the patients with NK/T cell lymphoma.

DETAILED DESCRIPTION:
Patients with NK/T cell lymphoma usually have a bad prognosis. These patients cannot be treated successfully with the conventional chemotherapy of CHOP.The investigators did this trial to evaluate the efficacy and tolerability of the combination chemotherapy of DICE in the patients with NK/T cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Age range 18-75 years old
* Histological confirmed NK/T cell lymphoma
* ECOG performance status less than 2
* Life expectancy of more than 3 months
* None of major drugs in the trial (IFO,VP16,DDP) has been previously used
* Normal laboratory values: hemoglobin > 80 g/dl, neutrophil > 2×109/L, platelet > 100×109/L, serum creatine < 1.5×upper limitation of normal (ULN), serum bilirubin < 1.5×ULN, ALT and AST < 2.5×ULN

Exclusion Criteria:

* Pregnant or lactating women
* Serious uncontrolled diseases and intercurrent infection
* The evidence of CNS metastasis
* History of other malignancies except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-03; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Response rate | every two cycles

SECONDARY OUTCOMES:
TTP and OS | every two cycles

CONTACTS AND LOCATIONS:
Overall Officials: Ye Guo, M.D., Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China